CLINICAL TRIAL: NCT02844972
Title: Interest of Pain Assessment by the Family of Patients in Limiting and Stopping Active Treatment Process Admitted in ER. Study DOFAMILA
Acronym: DOFAMILIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0216
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Patient's Pain in Later Life
Keywords: arrest or limitation of active treatment; emergency treatment
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Decisions to limit and stop active therapeutics are common in the emergency unit. They are framed by the Leonetti law of 22 April 2005 recommending the refusal of unreasonable obstinacy and care of the patient's pain in later life. The pain assessment is an issue for these patients whose in majority, are not communicating. Moreover, no specific tool and the teams in charge, not knowing the patient make the recognition and treatment of pain symptoms very complex. This is the potential interest of directly involving the family or the person of confidence in this management , the first step being the detection and evaluation of pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18
* non communicating patients admitted in emergency ward
* unanimous decision of stopping and limiting active treatment according to Leonetti's law of April 22nd, 2005
* Presence of a member of the patients family or one of his legal representative

Exclusion Criteria:

* Children
* no health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non communicating patients admitted in emergency ward
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
simplified verbal scale | admission time in ER (Day 1)
  A simplified verbal scale with 5 levels used by caregivers and family to evaluate the intensity of pain, "painless", "little sore", "moderately painful", "very painful", "extremely painful".
  Compare the pain assessment by the family or the person of trust and care teams within a population of non-communicating patients for whom a decision of limiting and stopping active treatment is taken emergency ward.

SECONDARY OUTCOMES:
simplified verbal scale | 24 hours after the decision of limiting or stopping active treatment in emergencies
  A simplified verbal scale with 5 levels used by caregivers and family to evaluate the intensity of pain, "painless", "little sore," "moderately painful", "very painful", "extremely painful ".
  Compare the pain assessment by the family or the person of trust and care teams within a population of non-communicating patients 24 hours after the decision of limiting or stopping active treatment in emergencies
Algoplus scale | at admission (Day 1)
  Comparison of pain assessment between families and caregivers with support will be made using Algoplus scale defining a pain when the score is greater than 2.
  Compare the pain assessment by the family or the person of trust and care teams with the support of a rating scale in a population of non-communicating patients for whom a decision of limiting or stopping active treatment in emergencies.
PAINAD scale | at admission (Day 1)
  Comparison of pain assessment between families and caregivers with support will be made using PAINAD scale rated from 0 to 10, defining the intensity of pain.
  Compare the pain assessment by the family or the person of trust and care teams with the support of a rating scale in a population of non-communicating patients for whom a decision of limiting or stopping active treatment in emergencies
CAESAR scale | 24 hours after admission
  Assess the feelings of nursing teams on the family involvement in the assessment of pain and not communicating patient discomfort for which is a determination of limiting or stopping active treatment in emergencies.
CAESAR scale | 3 weeks after admission
  The experience of the family will be described based on the questionnaire adapted from CAESAR scale ( rating scale of the quality of the care of the dying in intensive care) .
  Assess the feelings of nursing teams on the family involvement in the assessment of pain and not communicating patient discomfort for which is a determination of limiting or stopping active treatment in emergencies.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JACQUIN, MD, Principal Investigator — ER unit Hospital Edouard Herriot, Hospices Civils de Lyon
Locations (1):
- ER unit Hospital Edouard Herriot, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Douplat M, Daoud K, Berthiller J, Schott AM, Potinet V, Le Coz P, Tazarourte K, Jacquin L. Poor Involvement of General Practitioners in Decisions of Withholding or Withdrawing Life-Sustaining Treatment in Emergency Departments. J Gen Intern Med. 2020 Jan;35(1):177-181. doi: 10.1007/s11606-019-05464-y. Epub 2019 Nov 4. PMID 31686289